CLINICAL TRIAL: NCT00038610
Title: Phase II Study of Hyper-CVAD Plus Imatinib Mesylate (Gleevec, STI571) for Philadelphia-Positive Acute Lymphocytic Leukemia
Brief Title: Study of Hyper-CVAD Plus Imatinib Mesylate for Philadelphia-Positive Acute Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID01-006; NCI-2012-01487 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2002-06-03; First posted 2002-06-04 (Estimated); Results first posted 2015-09-18 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-08

CONDITIONS: Leukemia
Keywords: Leukemia; Lymphoblastic; Acute; Philadelphia-Positive; Imatinib Mesylate; Gleevec; Glivec; Imatinib; STI571; STI-571; CGP-57148B; NSC-716051; Cyclophosphamide; Cytoxan®,; Neosar®; Doxorubicin; Adriamycin ®; Rubex ®; Adriamycin PFS; Adriamycin RDF; Vincristine; Dexamethasone; Decadron; Methotrexate; Cytarabine; Ara-C; Cytosar; DepoCyt; Cytosine Arabinosine Hydrochloride; Mesna; Mesnex; G-CSF; Filgrastim; Neupogen
MeSH Terms: conditions — Leukemia | interventions — Imatinib Mesylate; Cyclophosphamide; Doxorubicin; Vincristine; Dexamethasone; Calcium Dobesilate; Methotrexate; Cytarabine; Mesna; Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hyper-CVAD + Imatinib (Experimental): Imatinib 600 mg orally days 1-14, course 1, & 600 mg daily days 1-14 (daily if tolerated course 1), even courses. Cyclophosphamide 300 mg/m^2 intravenous (IV) for 6 doses days 1-3, odd courses. Doxorubicin 50 mg/m^2 IV day 4; Vincristine 2 mg IV days 4 & 11; & Dexamethasone 40 mg IV or orally daily days 1-4 & 11-14 odd courses 1, 3, 5, 7. Methotrexate 12 mg intrathecally (6 mg if via Ommaya reservoir) day 2, odd courses and 200 mg/m^2 IV over 2 hours followed by 800 mg/m^2 over 22 hours day 1 of even courses. Cytarabine 100 mg intrathecally day 7 for odd courses and 3 gm/m^2 IV every 12 hours for 4 doses days 2-3 for even courses. Mesna 600 mg/m^2 IV daily, odd courses. G-CSF 10 mcg/kg/day after completion of chemotherapy until neutrophil recovery to 1 x 109/L or higher for all courses.
  Interventions: Drug: Imatinib Mesylate; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Dexamethasone; Drug: Methotrexate; Drug: Cytarabine; Drug: Mesna; Drug: G-CSF

INTERVENTIONS:
Drug: Imatinib Mesylate — 600 mg by mouth on days 1 - 14 for course 1, and 600 mg by mouth daily days 1-14 (or daily if tolerated with course 1) for courses 2, 4, 6, 8.
  Other Names: Gleevec; Glivec; Imatinib; STI571; STI-571; CGP-57148B; NSC-716051
Drug: Cyclophosphamide — 300 mg/m^2 by vein every 12 hours for 6 doses days 1, 2, 3 (total dose 1800 mg/m^2) for courses 1, 3, 5, 7.
  Other Names: Cytoxan®,; Neosar®
Drug: Doxorubicin — 50 mg/m^2 by vein on day 4 after last dose of CTX for courses 1, 3, 5, 7.
  Other Names: Adriamycin ®; Rubex ®; Adriamycin PFS; Adriamycin RDF
Drug: Vincristine — 2 mg by vein on day 4 and day 11 for courses 1, 3, 5, 7.
Drug: Dexamethasone — 40 mg by vein or by mouth daily on days 1 - 4 and days 11 - 14 for courses 1, 3, 5, 7.
  Other Names: Decadron
Drug: Methotrexate — 12 mg intrathecally (6 mg if via Ommaya reservoir) day 2 for courses 1, 3, 5, 7.
  200 mg/m^2 by vein over 2 hours followed by 800 mg/m^2 over 22 hours on day 1 of courses 2, 4, 6, 8.
Drug: Cytarabine — 100 mg intrathecally day 7 for courses 1, 3, 5, 7.
  3 gm/m2 by vein over 2 hrs every 12 hrs for 4 doses on days 2 and 3 for courses 2, 4, 6, 8.
  Other Names: Ara-C; Cytosar; DepoCyt; Cytosine Arabinosine Hydrochloride
Drug: Mesna — 600 mg/m^2 by vein daily for 24 hours for courses 1, 3, 5, 7.
  Other Names: Mesnex
Drug: G-CSF — 10 mcg/kg/day after completion of chemotherapy until neutrophil recovery to 1 x 109/L or higher for all courses.
  Other Names: Filgrastim; Neupogen

SUMMARY:
The goal of this clinical research study is to learn if intensive chemotherapy, combined with imatinib mesylate (Gleevec, STI571) given for 8 courses over 6 months, followed by maintenance imatinib mesylate plus chemotherapy for 2 years, followed by imatinib mesylate indefinitely can improve Philadelphia-positive acute lymphoblastic leukemia. The safety of this treatment will also be studied.

DETAILED DESCRIPTION:
Before treatment starts, patients will have a complete exam, including medical history and documentation of disease, blood, and marrow tests. A chest x-ray will be taken. CT scans may be taken if needed. A bone marrow sample will be taken through a large needle. An EKG and MUGA (heart function tests) will be performed.

During treatment, patients will give blood samples (about 1 tablespoon each) at least twice a week. A bone marrow sample will be repeated 2 and 3 weeks from the beginning of treatment to check on response. After two courses of chemotherapy, the tests done before treatment will be repeated to check for response.

All patients will receive 2 kinds of chemotherapy courses for a total of 8 courses. Chemotherapy courses will be given through a large vein by a central venous catheter (a plastic tube usually placed under the collarbone). Imatinib mesylate will be given as a pill with the chemotherapy.

Course 1 will start with cyclophosphamide given by vein over 2-3 hours every 12 hours for 6 doses over 3 days (Days 1,2,3). Mesna will be given by vein continuously for 4 days with the cyclophosphamide to protect the bladder. Doxorubicin will be given by vein over 24 hours on Day 4. Vincristine will be given by short infusion on Days 4 and 11. Dexamethasone (a steroid) will be given by mouth or by vein on Days 1-4 and 11-14. The imatinib mesylate will be given by mouth with breakfast and a large glass of water daily on Days 1-14. Medicines will be given to prevent nausea and to protect the kidneys from increased amounts of uric acid, which may be released when leukemia cells die.

G-CSF (growth stimulating colony factor) will be given after completion of the chemotherapy. It is given to allow for rapid recovery of the normal marrow. G-CSF will be injected under the skin until the counts recover. Treatment to the brain will be given inside the spinal fluid with methotrexate around Day 2 and cytarabine about day 7. This is done to prevent the leukemia from developing there.

For patients aged 60 years or older, this Course 1 will be given in a protective isolation room to decrease the risk of infection(s).

During Course 2, patients will be given methotrexate by infusion over 24 hours on the first day and cytarabine at a high dose over 2 hours every 12 hours for 4 doses (Days 2 and 3). Citrovorum factor (leucovorin), an antidote for side effects of methotrexate, will be given by vein or by mouth for 2-3 days (Day 2 and on). Solumedrol (a steroid) will be given by vein every 12 hours for 6 doses. Imatinib mesylate will be given by mouth with breakfast and a large glass of water on Days 1-14 or daily, depending on tolerance with Course 1. G-CSF will be given as in Course 1. The treatment to the brain inside the spinal fluid will be given as in Course 1 around Days 2 and 7.

The chemotherapy will alternate between hyper-CVAD plus imatinib mesylate (Courses 1, 3, 5, and 7) and methotrexate/cytarabine plus imatinib mesylate (Courses 2, 4, 6, and 8) to complete a total of 8 courses. G-CSF will be given as in Course 1. Anti-nausea medicine will be given with each course of chemotherapy. The urine will be alkalized to protect the kidneys. Antibiotics will be given by mouth to prevent infection.

After the 8 courses, monthly maintenance chemotherapy plus imatinib mesylate will be given. This includes daily imatinib mesylate, monthly vincristine by vein, and prednisone by mouth for 5 days every month. Maintenance chemotherapy will be given for a total of 24 months, and will be interrupted by 2 periods of intensive chemotherapy courses with hyper-CVAD and imatinib mesylate at 6 and 13 months from the start of maintenance. Imatinib mesylate will be continued daily as tolerated indefinitely.

After two courses of the intensive chemotherapy, the response to the treatment will be evaluated. If the leukemia is responding, the therapy will be continued. Patients will be taken off study if the leukemia starts to get worse.

During and after completion of treatment, patients will have a complete exam, including blood tests. If needed, a chest X-ray or CT scan will be done. A bone marrow sample will be taken through a large needle. Patients will then return every 2 to 3 months for a checkup, including blood and bone marrow. X-rays and heart studies (MUGA or ECG) may be repeated if needed.

An Ommaya reservoir may also be placed surgically as a route to treat leukemia in the brain or to prevent leukemia in patients who have difficulty with the spinal treatments. An Ommaya reservoir is an access port inserted under the skin of the scalp that enters into the spinal fluid cavity of the brain.

Treatment will be given on an inpatient basis (3 to 5 days) for the 8 intensive courses of chemotherapy, or as indicated by the clinical condition. The maintenance treatments will be given as an outpatient, except for the courses of hyper-CVAD and imatinib mesylate.

This is an investigational study. The FDA has approved imatinib mesylate for use in chronic myelogenous leukemia and other clinical research studies. About 55 patients will take part in this study. All will be from MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of previously untreated Ph-positive ALL or previously treated in CR after 1-2 courses of therapy or failure after one course of induction chemotherapy without imatinib mesylate.
2. Age > or = 15 years. Those < 15 years of age will be treated under compassionate IND.
3. Zubrod performance status < or = 2 (ECOG Scale, Appendix A).
4. Adequate liver function (bilirubin < or = to 3.0 mg/dl, unless considered due to tumor), and renal function (creatinine < or = to 3.0 mg/dl, unless considered due to tumor).
5. Adequate cardiac function as assessed clinically by physical examination.
6. Signed informed consent.

Exclusion Criteria:

1. Active serious infection not controlled by oral or intravenous antibiotics.
2. Treatment with investigational antileukemic agent or chemotherapy agents in the last 7 days before study entry, unless full recovery from side-effects has occurred or patient has rapidly progressive disease judged life-threatening.
3. Active secondary malignancy other than skin cancer (e.g. basal cell carcinoma or squamous cell carcinoma) than in investigator's opinion will shorten survival to less than 1 year.
4. History of Grade III/IV cardiac problems as defined by the New York Heart Association Criteria.
5. Prior history of treatment with imatinib mesylate.
6. Pregnancy or lactating in women of childbearing potential.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2001-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naval Daver, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Ribera JM, Prawitz T, Freitag A, Sharma A, Dobi B, Rizzo F, Sabatelli L, Patos P. Ponatinib vs. Imatinib as Frontline Treatment for Philadelphia Chromosome-Positive Acute Lymphoblastic Leukemia: A Matching Adjusted Indirect Comparison. Adv Ther. 2023 Jul;40(7):3087-3103. doi: 10.1007/s12325-023-02497-y. Epub 2023 May 19. PMID 37208556
- [Derived] Daver N, Thomas D, Ravandi F, Cortes J, Garris R, Jabbour E, Garcia-Manero G, Borthakur G, Kadia T, Rytting M, Konopleva M, Kantarjian H, O'Brien S. Final report of a phase II study of imatinib mesylate with hyper-CVAD for the front-line treatment of adult patients with Philadelphia chromosome-positive acute lymphoblastic leukemia. Haematologica. 2015 May;100(5):653-61. doi: 10.3324/haematol.2014.118588. Epub 2015 Feb 14. PMID 25682595
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: March 28, 2001 to October 04, 2006. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | Hyper-CVAD + Imatinib
Started | 54
Completed | 54
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Hyper-CVAD + Imatinib
Number analyzed (Participants) | 54
Age, Continuous [Median (Full Range); unit: years] | 51 [17 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 28
Region of Enrollment [Number; unit: participants]
  United States | 54

OUTCOME MEASURES:

1. Primary Outcome: Response To Induction Therapy With Hyper-CVAD Plus Imatinib Mesylate
Description: Complete Remission (CR): Defined as the presence of 5% or less blasts in the bone marrow, with a granulocyte count of 1.0 × 109/L or higher and a platelet count of 100 × 109/L and no extramedullary disease.
  Partial Response (PR): As above for CR except for the presence of 6-25% marrow blasts.
  Molecular CR: Same as for CR with RT-PCR negativity for bcr-abl.
  Induction Death: Defined as death occurring after start of therapy without meeting the definition of CR or resistant disease.
Time Frame: Baseline to 6 months
Population: Of the 54 participants, 39 (72%) presented with de novo disease, 6 (11%) were refractory to standard induction therapy, and 9 (17%) entered the study in complete remission (CR) after one course of standard induction therapy.
Measure: Number; unit: participants
Arm/Group | Hyper-CVAD + Imatinib
Number analyzed (Participants) | 54
participants
  Complete Remission | 42
  Partial Remission | 1
  Molecular Complete Remission | 17
  Induction Death | 1

2. Secondary Outcome: Overall Survival Rate at 2-year and 5-year.
Description: Overall survival (OS) was calculated from the date of initiation of therapy until death.
Time Frame: Baseline to 2-year and 5-year
Measure: Number; unit: percentage of participants
Arm/Group | Hyper-CVAD + Imatinib
Number analyzed (Participants) | 54
percentage of participants
  2-year OS rate | 57
  5-year OS rate | 43

3. Primary Outcome: Disease-Free Survival Rate at 2-year and 5-year.
Description: Disease-Free Survival (DFS) was calculated from the time of complete remission until relapse or death due to any cause.
Time Frame: Baseline to 2-year and 5-year
Measure: Number; unit: percentage of participants
Arm/Group | Hyper-CVAD + Imatinib
Number analyzed (Participants) | 54
percentage of participants
  2-year DFS rate | 49
  5-year DFS rate | 43

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were collected from receiving of induction therapy to discontinuation of study drug. Collection period: April, 2001 to June 2013.
Arm/Group | Hyper-CVAD + Imatinib
Serious Adverse Events (participants affected / at risk) | 36/54
Other Adverse Events (participants affected / at risk) | 54/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hyper-CVAD + Imatinib (N=54)
Pericardial and pleural effusion (Cardiac disorders) | 1 (1)
Death (General disorders) | 35 (35)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hyper-CVAD + Imatinib (N=54)
ALBUMIN, SERUM-LOW (Metabolism and nutrition disorders) | 1 (1)
BILIRUBIN INCREASE (Metabolism and nutrition disorders) | 2 (3)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 3 (3)
CONSTIPATION (Gastrointestinal disorders) | 2 (3)
DEHYDRATION (Gastrointestinal disorders) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 3 (4)
DIZZINESS (Nervous system disorders) | 1 (2)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 3 (4)
DYSRHYTHMIA (Cardiac disorders) | 1 (1)
EDEMA (Blood and lymphatic system disorders) | 6 (8)
FATIGUE (General disorders) | 3 (3)
FEVER NEUTROPENIC (Infections and infestations) | 7 (13)
FEVER WITHOUT NEUTROPENIA (General disorders) | 3 (4)
GASTRITIS (Gastrointestinal disorders) | 2 (2)
GLUCOSE, SERUM-HIGH (Metabolism and nutrition disorders) | 4 (5)
HEADACHE (Nervous system disorders) | 6 (7)
HEMORRHOIDAL BLEED (Gastrointestinal disorders) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 1 (2)
HYPOKALEMIA (Metabolism and nutrition disorders) | 3 (4)
HYPONATREMIA (Metabolism and nutrition disorders) | 2 (2)
HYPOTENSION (Cardiac disorders) | 1 (2)
INFECTION FEBRILE NEUTROPENIA (Infections and infestations) | 5 (6)
INFECTION NEUTROPENIC (Infections and infestations) | 2 (3)
INFECTION WITHOUT NEUTROPENIA (Infections and infestations) | 3 (4)
MOTOR (Musculoskeletal and connective tissue disorders) | 1 (1)
NAUSEA ALONE (Gastrointestinal disorders) | 6 (7)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PLEURITIC PAIN (General disorders) | 1 (2)
PRURITUS/ITCHING (Skin and subcutaneous tissue disorders) | 2 (3)
RENAL GENITOURINARY (Renal and urinary disorders) | 1 (1)
WOUND INFECTION (Infections and infestations) | 2 (2)
URINARY TRACT INFECTION (Renal and urinary disorders) | 1 (1)
INFECTION (Infections and infestations) | 4 (5)
SENSORY (Nervous system disorders) | 3 (3)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
TACHYCARDIA (Cardiac disorders) | 1 (1)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 2 (2)
SYNCOPE (Nervous system disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 4 (4)
STOMATITIS (Gastrointestinal disorders) | 1 (4)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 2 (2)
TRANSAMINASE INCREASE (Metabolism and nutrition disorders) | 1 (1)
THROMBOSIS/EMBOLISM (Vascular disorders) | 3 (3)
EPISTAXIS (General disorders) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 1 (1)
SPEECH IMPAIRMENT (Nervous system disorders) | 1 (1)
CREATININE INCREASE (Metabolism and nutrition disorders) | 2 (2)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
FIBRINOGEN DECREASE (Metabolism and nutrition disorders) | 1 (1)
FRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1)
CARDIAC (Cardiac disorders) | 1 (1)
BACK PAIN (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes